CLINICAL TRIAL: NCT04761302
Title: Postoperative Pain Management in Patients Undergoing Intramedullary Nail Fixation After Tibia and Femoral Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A9290220
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Femur Fracture; Tibial Fractures
Keywords: Opioid use; Post-operative pain; Analgesic use; Femur fracture; Tibia fracture; Intramedullary Nailing
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures; Pain, Postoperative | interventions — Acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and oral acetaminophen (Experimental): Group 1 will be composed of tibial fracture patients receiving the following standard pain control protocol: ketorolac 30 mg intravenous (IV) every 6 hours for patients younger than 70 years versus ketorolac 15 mg IV every 6 hours for patients older than 70 years, first dose will be administered 30 minutes preoperatively. An additional 1000mg of oral acetaminophen will be administered every 6 hours simultaneously regardless of the age group. Patients who determine pain to be unbearable and wish to opt out of the non-opioid group will receive may do so.
  Interventions: Drug: Intravenous ketorolac and oral acetaminophen
- Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and oral oxycodone (Active Comparator): Group 2 will be composed of tibial fracture patients receiving the following pain control protocol: morphine 0.1 mg per kg intravenous every 6 hours with an additional oral oxycodone combined with acetaminophen 2 tabs every 6 hours.
  Interventions: Drug: Intravenous morphine and oral oxycodone
- Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen (Experimental): Group 3 will be composed of femoral fracture patients receiving the following standard pain control protocol: ketorolac 30 mg intravenous (IV) every 6 hours for patients younger than 70 years versus ketorolac 15 mg IV every 6 hours for patients older than 70 years, first dose will be administered 30 minutes preoperatively. An additional 1000mg of oral acetaminophen will be administered every 6 hours simultaneously regardless of the age group. Patients who determine pain to be unbearable and wish to opt out of the non-opioid group will receive may do so.
  Interventions: Drug: Intravenous ketorolac and oral acetaminophen
- Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and oral oxycodone (Active Comparator): Group 4 will be composed of femoral fracture patients receiving the following pain control protocol: morphine 0.1 mg per kg intravenous every 6 hours with an additional oral oxycodone combined with acetaminophen 2 tabs every 6 hours.
  Interventions: Drug: Intravenous morphine and oral oxycodone

INTERVENTIONS:
Drug: Intravenous ketorolac and oral acetaminophen — ketorolac 30 mg intravenous (IV) every 6 hours for patients younger than 70 years versus ketorolac 15 mg IV every 6 hours for patients older than 70 years, first dose will be administered 30 minutes preoperatively. An additional 1000mg of oral acetaminophen will be administered every 6 hours simultaneously regardless of the age group
  Arms: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and oral acetaminophen; Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen
Drug: Intravenous morphine and oral oxycodone — Morphine 0.1 mg per kg intravenous every 6 hours with an additional oral oxycodone combined with acetaminophen 2 tabs every 6 hours.
  Arms: Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and oral oxycodone; Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and oral oxycodone

SUMMARY:
The purpose of this trial is to determine whether oral acetaminophen and intravenous ketorolac are viable alternatives to opioid medication regimens for the pain management of patients with tibial and femoral shaft fractures treated with intramedullary nailing. This study will explore an alternative for opioid medications for patients undergoing intramedullary nailing of tibial and femoral shaft fractures.

DETAILED DESCRIPTION:
The data analysis for the study will be performed separately for patients with femoral fractures and for patients with tibial fractures. Therefore, the data analysis will compare patients with femoral fractures receiving the experimental treatment to patients with femoral fractures receiving the control treatment (Group 1 vs. Group 2). Likewise, patients with tibial fractures receiving the experimental treatment will be compared to patients with tibial fractures receiving the control treatment (Group 3 vs. Group 4).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with tibial and femoral shaft fractures
2. Patients undergoing intramedullary nailing
3. Willing to participate in the protocol

Exclusion Criteria:

1. Chronic pain disorder (daily use of oral opioids)
2. Allergy or hypersensitivity to non steroid anti-inflammatory drug
3. Impaired renal, cardiac, or hepatic function
4. History of gastrointestinal bleeding or substance abuse

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis F. Lojo-Sojo, MD, Principal Investigator — Orthopaedic Surgery Section, University of Puerto Rico Medical Sciences Campus San Juan, Puerto Rico
Locations (1):
- University District Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess-Arcelay H, Claudio-Marcano A, Torres-Lugo NJ, Deliz-Jimenez D, Acosta-Julbe J, Hernandez G, Deliz-Jimenez D, Monge G, Ramirez N, Lojo-Sojo L. Opioid-Sparing Nonsteroid Anti-inflammatory Drugs Protocol in Patients Undergoing Intramedullary Nailing of Tibial Shaft Fractures: A Randomized Control Trial. J Am Acad Orthop Surg. 2024 Jun 15;32(12):e596-e604. doi: 10.5435/JAAOS-D-23-01014. Epub 2024 Apr 4. PMID 38579315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Started | 52 | 44 | 29 | 42
Completed | 52 | 44 | 29 | 42
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone: Group 4 will be composed of tibial fracture patients receiving the following pain control protocol: morphine 0.1 mg per kg intravenous every 6 hours with an additional oral oxycodone combined with acetaminophen 2 tabs every 6 hours.
- Total: Total of all reporting groups
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Total
Number analyzed (Participants) | 52 | 44 | 29 | 42 | 167
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 31 [23 to 42] | 40 [27 to 60] | 31 [23 to 42] | 40 [27 to 60] | 36 [24 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 6 | 13 | 36
  Male | 45 | 34 | 23 | 29 | 131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 26.6 (5.90) | 26.9 (6.21) | 27.1 (7.1) | 26.7 (6.2) | 26.8 (6.3)
Smoker status [Count of Participants; unit: Participants]
  Smoker | 13 | 12 | 6 | 13 | 44
  Non-smoker | 39 | 32 | 23 | 29 | 123
Diabetes Status [Count of Participants; unit: Participants]
  Yes | 5 | 5 | 3 | 8 | 21
  No | 47 | 39 | 26 | 34 | 146

OUTCOME MEASURES:

1. Primary Outcome: 12hrs VAS Pain Scores
Description: Visual Analog Scale; 0-10 (10 indicates highest degree of pain)
Time Frame: Measured at postoperative hour 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone: Group 2 will be composed of tibial fracture patients receiving the following pain control protocol: morphine 0.1 mg per kg intravenous every 6 hours with an additional oral oxycodone combined with acetaminophen 2 tabs every 6 hours.
  Use of non-steroid anti-inflammatory drugs (NSAIDS) as an alternative for post-operative pain management after a femur and tibia fracture: This is a randomized controlled, single blind, parallel groups, opioid control trial of all patients (total of 150 patients) who suffered tibial and femoral shaft fractures and were treated with intramedullary nailing. Patients will be aleatory assigned to two study groups: Group-1 will receive non-opioid medications, and Group-2 will receive opioid medications. During the inpatient postoperative period, patients will undergo subjective evaluation of pain utilizing a previously validated questionnaire, the Visual Analogue Score (VAS). The first questionnaire will be completed twelve hours after surgery and during subsequent twelve-hour intervals until discharge. Secondary outcomes will include efficiency such as time to gastrointestinal motility, time to weight bearing of affected limb, resumption of ambulation, and length of hospital stay. The evaluation will take approximately 15 minutes to complete each time, we the entire participation time to be 60 minutes.
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
score on a scale | 7.6 (2.20) | 7.9 (2.01) | 7.3 (2.5) | 7.2 (2.0)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.215, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.445, t-test, 2 sided — A priori threshold for statistical significance: <0.05

2. Primary Outcome: 24hrs VAS Pain Score
Description: Visual Analog Scale; 0 to 10 (10 indicates highest degree of pain)
Time Frame: Measured at postoperative hour 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
score on a scale | 4.9 (2.5) | 5.9 (2.6) | 5.4 (2.6) | 5.1 (2.4)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.041, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.300, t-test, 2 sided — A priori threshold for statistical significance: <0.05

3. Primary Outcome: 36hrs VAS Pain Scores
Description: Visual Analog Scale; 0-10 (10 indicates highest degree of pain)
Time Frame: Measured at postoperative hour 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
score on a scale | 4.9 (2.5) | 5.63 (2.3) | 5.3 (1.8) | 5.6 (2.3)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.12, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.359, t-test, 2 sided — A priori threshold for statistical significance: <0.05

4. Primary Outcome: 48hrs VAS Pain Scores
Description: Visual Analog Scale; 0-10 (10 indicates highest degree of pain)
Time Frame: Measured at postoperative hour 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
score on a scale | 3.6 (2.01) | 4.3 (2.6) | 4.0 (1.6) | 3.4 (2.2)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.083, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.152, t-test, 2 sided — A priori threshold for statistical significance: <0.05

5. Primary Outcome: 12hrs MME
Description: Opioid consumption at postoperative hour 12. Reported as Morphine Milligram Equivalents (MME)
Time Frame: Measured at postoperative hour 12
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
Morphine Milligram Equivalents (MME) | 2.9 (7.5) | 8.5 (10.1) | 2.9 (4.5) | 12.1 (11.6)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.002, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priori threshold for statistical significance: <0.05

6. Primary Outcome: 24hrs MME
Description: Opioid consumption at postoperative hour 24. Reported as Morphine Milligram Equivalents (MME)
Time Frame: Measured at postoperative hour 24
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
Morphine Milligram Equivalents (MME) | 9.2 (18.6) | 21.49 (22.4) | 10.4 (13.6) | 28.8 (20.6)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.002, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priori threshold for statistical significance: <0.05

7. Primary Outcome: 36hrs MME
Description: Opioid consumption at postoperative hour 36. Reported as Morphine Milligram Equivalents (MME)
Time Frame: Measured at postoperative hour 36
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
Morphine Milligram Equivalents (MME) | 14.1 (25.9) | 29.5 (29.9) | 15.7 (15.9) | 36.6 (29.1)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.004, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priori threshold for statistical significance: <0.05

8. Primary Outcome: 48hrs MME
Description: Opioid consumption at postoperative hour 48. Reported as Morphine Milligram Equivalents (MME)
Time Frame: Measured at postoperative hour 48
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
Morphine Milligram Equivalents (MME) | 18.3 (33.3) | 37.2 (37.8) | 20.1 (21.0) | 48.0 (35.6)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.006, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priori threshold for statistical significance: <0.05

9. Secondary Outcome: Hospital Length of Stay
Description: Time from intervention to discharge
Time Frame: Determined by discharge date
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
Number analyzed (Participants) | 52 | 44 | 29 | 42
Days | 1.9 (0.61) | 2.00 (0.89) | 1.8 (0.5) | 1.9 (1.1)
Statistical Analysis 1: Comparison: Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.354, t-test, 2 sided — A priori threshold for statistical significance: <0.05
Statistical Analysis 2: Comparison: Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen vs Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone; Test type: Superiority; p = 0.455, t-test, 2 sided — A priori threshold for statistical significance: <0.05

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/46 | 0/29 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/52 | 3/46 | 7/29 | 8/42
Other Adverse Events (participants affected / at risk) | 0/52 | 0/46 | 0/29 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Tibial Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen (N=52) | Group 2: Tibial Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone (N=46) | Group 3: Femoral Fracture Patients Receiving Intravenous Ketorolac and Oral Acetaminophen (N=29) | Group 4: Femoral Fracture Patients Receiving Intravenous Morphine and Oral Oxycodone (N=42)
Non-Union (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 — Non-Union was defined as a delayed union that did not resolve at 9 months after surgery.
Delayed Union (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 6 — Delayed union was defined as a lack of callous formation at 6 months after surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT04761302/Prot_SAP_004.pdf
  • Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT04761302/ICF_005.pdf